CLINICAL TRIAL: NCT06742515
Title: Blinatumomab Combined With Reduced-dose Chemotherapy in Treating Precursor B Cell Acute Lymphoblastic Leukemia: a Phase II, Single Arm and Multicenter Study
Brief Title: Blinatumomab Plus Reduced-dose Chemotherapy in Treating B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240126C
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-09

CONDITIONS: Precursor B-Cell Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Blinatumomab plus Reduced-dose Chemotherapy
  Interventions: Drug: Blinatumomab plus Reduced-dose Chemotherapy

INTERVENTIONS:
Drug: Blinatumomab plus Reduced-dose Chemotherapy — Cycle 1: Reduced VCP on day1, IV and Blinatumomab for 2 weeks, IV. Cycle 2: Blinatumomab for 2 weeks, IV and Venetoclax for 2 weeks, oral.

SUMMARY:
Precursor B cell acute lymphoblastic leukemia (B-ALL) is an aggressive type of leukemia, with high relapse rate and poor long term survival in adults. Traditional treatment regimens mainly include chemotherapy and hematopoietic stem cell transplantation. In the past decade, with the application of molecular targeted drugs and immunotherapy, the survival of B-ALL patients has significantly improved. In this study，we propose a treatment approach that combines Blinatumomab and Reduced-dose Chemotherapy in B-ALL adults. Our study aims to answer the safety and efficacy of this treatment regimen, and further improve the survival for those participants.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II and open-label study. A total of 20 Ph-negative B-ALL participants will be enrolled. The primary endpoint is MRD-negative CR rate. The induction therapy is a combination of Blinatumomab(Blina), Vindesine(VDS), Cyclophosphamide(CTX) and Dexamethasone(DXM). The second cycle would be the combination of Blina and Venetoclax(VEN). As for consolidation therapy, we suggest the bone marrow transplantation. The purpose of this study is to explore the safety and efficacy of the treatment regimen in the treatment of newly diagnosed young Ph-negative B-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Before enrollment, patients must be diagnosed with de novo precursor B-cell acute lymphoblastic leukemia and be negative for Philadelphia chromosome. The diagnostic criteria refer to the 2022 WHO classification; 2. Age≥15 years， ≤59 years; 3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2; 4. Expected survival time ≥ 2 months; 5. No organ dysfunction that would restrict the use of this protocol during the screening period; 6. Understand the study and sign the informed consent form. 7. Men, women of childbearing age (only postmenopausal women who have been menopausal for at least 12 months can be considered infertile), and their partners voluntarily take effective contraceptive measures deemed effective by the investigator during the treatment period and for at least 12 months after the last dose of the study drug.

Exclusion Criteria:

* 1. Patients with known central nervous system (CNS) involvement of ALL; 2. Diseases with abnormal heart, lung, liver, kidney, or other organ functions that may limit the patient's participation in this trial (including but not limited to severe infections, uncontrolled diabetes, severe heart failure or angina, active pulmonary tuberculosis, asthma, COPD, bronchiectasis, etc.); 3. Cardiac ultrasound LVEF < 45%; 4. History of other malignancies within the past 5 years, excluding localized thyroid cancer and in situ skin cancer; 5. Serum total bilirubin > 1.5 ULN (upper limit of normal); ALT or AST > 2.5 ULN; serum creatinine > 1.5 ULN; 6. Known HIV infection; 7. Conditions affecting the use of the study drug as assessed by the investigator; 8. Unable to understand or comply with the study protocol.

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate with negative minimal residual disease | at the end of cycle 1 and 2（each cycle is 28 days）
  complete remission and negative MRD detected by flowcytometry

SECONDARY OUTCOMES:
CR/CRi after Cycle 1 and 2 | at the end of cycle 1 and 2（each cycle is 28 days）
  Blast rate lower than 5% with or without peripheral blood cell recovery
Minimal residual disease(MRD) | At the end of each cycle（each cycle is 28 days）
  MRD level detected by flow cytometry which value <0.1% is defined as negtive
Overall survival (OS) | up to 5 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of death from any cause;
Event free survival(EFS) | up to 5 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first;

OTHER OUTCOMES:
Minimal residual disease (MRD) | At the end of Cycle 1 and 2（each cycle is 28 days）
  MRD level detected by next generation sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang 310003, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Open in the form of original data report before December 30, 2028
Supporting Information: CSR

REFERENCES:
- [Background] Beldjord K, Chevret S, Asnafi V, Huguet F, Boulland ML, Leguay T, Thomas X, Cayuela JM, Grardel N, Chalandon Y, Boissel N, Schaefer B, Delabesse E, Cave H, Chevallier P, Buzyn A, Fest T, Reman O, Vernant JP, Lheritier V, Bene MC, Lafage M, Macintyre E, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Oncogenetics and minimal residual disease are independent outcome predictors in adult patients with acute lymphoblastic leukemia. Blood. 2014 Jun 12;123(24):3739-49. doi: 10.1182/blood-2014-01-547695. Epub 2014 Apr 16. PMID 24740809
- [Background] Lu J, Zhou H, Zhou X, Yang Y, Tong L, Miao M, Yang X, Chen S. Reduced-dose chemotherapy followed by blinatumomab in induction therapy for newly diagnosed B-cell acute lymphoblastic leukemia. Cancer Med. 2024 Mar;13(5):e7062. doi: 10.1002/cam4.7062. PMID 38491815
- [Background] Jabbour E, Short NJ, Senapati J, Jain N, Huang X, Daver N, DiNardo CD, Pemmaraju N, Wierda W, Garcia-Manero G, Montalban Bravo G, Sasaki K, Kadia TM, Khoury J, Wang SA, Haddad FG, Jacob J, Garris R, Ravandi F, Kantarjian HM. Mini-hyper-CVD plus inotuzumab ozogamicin, with or without blinatumomab, in the subgroup of older patients with newly diagnosed Philadelphia chromosome-negative B-cell acute lymphocytic leukaemia: long-term results of an open-label phase 2 trial. Lancet Haematol. 2023 Jun;10(6):e433-e444. doi: 10.1016/S2352-3026(23)00073-X. Epub 2023 May 12. PMID 37187201
- [Background] Litzow MR, Sun Z, Mattison RJ, Paietta EM, Roberts KG, Zhang Y, Racevskis J, Lazarus HM, Rowe JM, Arber DA, Wieduwilt MJ, Liedtke M, Bergeron J, Wood BL, Zhao Y, Wu G, Chang TC, Zhang W, Pratz KW, Dinner SN, Frey N, Gore SD, Bhatnagar B, Atallah EL, Uy GL, Jeyakumar D, Lin TL, Willman CL, DeAngelo DJ, Patel SB, Elliott MA, Advani AS, Tzachanis D, Vachhani P, Bhave RR, Sharon E, Little RF, Erba HP, Stone RM, Luger SM, Mullighan CG, Tallman MS. Blinatumomab for MRD-Negative Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2024 Jul 25;391(4):320-333. doi: 10.1056/NEJMoa2312948. PMID 39047240
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] Kantarjian H, Thomas D, O'Brien S, Cortes J, Giles F, Jeha S, Bueso-Ramos CE, Pierce S, Shan J, Koller C, Beran M, Keating M, Freireich EJ. Long-term follow-up results of hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone (Hyper-CVAD), a dose-intensive regimen, in adult acute lymphocytic leukemia. Cancer. 2004 Dec 15;101(12):2788-801. doi: 10.1002/cncr.20668. PMID 15481055
- [Background] Larson RA, Dodge RK, Burns CP, Lee EJ, Stone RM, Schulman P, Duggan D, Davey FR, Sobol RE, Frankel SR, et al. A five-drug remission induction regimen with intensive consolidation for adults with acute lymphoblastic leukemia: cancer and leukemia group B study 8811. Blood. 1995 Apr 15;85(8):2025-37. PMID 7718875
- [Background] Stock W, La M, Sanford B, Bloomfield CD, Vardiman JW, Gaynon P, Larson RA, Nachman J; Children's Cancer Group; Cancer and Leukemia Group B studies. What determines the outcomes for adolescents and young adults with acute lymphoblastic leukemia treated on cooperative group protocols? A comparison of Children's Cancer Group and Cancer and Leukemia Group B studies. Blood. 2008 Sep 1;112(5):1646-54. doi: 10.1182/blood-2008-01-130237. Epub 2008 May 23. PMID 18502832
- [Background] Jabbour EJ, Faderl S, Kantarjian HM. Adult acute lymphoblastic leukemia. Mayo Clin Proc. 2005 Nov;80(11):1517-27. doi: 10.4065/80.11.1517. PMID 16295033